CLINICAL TRIAL: NCT06229964
Title: A Double Blinded Randomized Controlled Trial (RCT) Exploring the Additional Effect of a Suprascapular Nerve Block in Combination with an Intra-Articular Corticosteroid Injection in Patients with Frozen Shoulder
Brief Title: Frozen Shoulder Treatment with Intra-Articular Corticosteroid Injection and Suprascapular Nerve Block
Acronym: FROSTBLOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23454_FROSTBLOCK
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Frozen Shoulder; Adhesive Capsulitis
Keywords: Frozen Shoulder; Adhesive Capsulitis of the Shoulder; Intra-articular corticosteroid injection; ultra-sound guided injection; suprascapular nerve block; Joint Diseases; Musculoskeletal Diseases; Bursitis
MeSH Terms: conditions — Bursitis; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective single-center Randomized Parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients will receive 2 concomitant USG injections: first a SSNB than an IACA Control group : short-acting SSNB is performed with a short-acting local anesthetic (Linisol 2%).
  Intervention group : SSNB is performed with a long-acting anesthestic (Ropivacaine 2%) + 20-mg methylprednisolone acetate.
  Same injected volume (5ml) in sham and intervention group. The advantage of using a short-acting anesthetic as a sham injection instead of a saline, is that at the time of injection the patient may perceive the anticipated short effect of the anesthetic similar to the intervention SSNB.
  The care provider will be unaware of the type of SSNB of the allocation group. The outcomes assessor will be unaware of the type of SSNB of the allocation group.
  The investigator who administers the injections, will be unaware of the allocation.
  The investigational products will be prepared by the pharmacist according to a pre-defined co-variate constrained randomization key.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SSNB + IACI (Active Comparator): Patients randomized to this arm will receive a SSNB (20-mg methylprednisolone acetate and 5-mL Ropivacaine 2mg/ml) than a IACI (40-mg methylprednisolone acetate and 1-mL Ropivacaine 2mg/ml).
  Rehabilitation/physiotherapy is considered standard of care.
  Interventions: Other: SSNB + IACI
- Short-acting SSNB + IACI (Placebo Comparator): Patients randomized to this arm will receive a SSNB (5-mL Linisol 10mg/ml) than a IACI (40-mg methylprednisolone acetate and 1-mL Ropivacaine 2mg/ml)
  Rehabilitation/physiotherapy is considered standard of care.
  Interventions: Other: Sham SSNB + IACI

INTERVENTIONS:
Other: SSNB + IACI — Usual care: All patients complete rehabilitation under supervision of their own physiotherapist. The investigators will provide some guidelines and criteria but is the physiotherapist's choice how to implement these guidelines in clinical practice.
  Patient education on home-exercises Monitoring of peak pain, at rest/night and after rehabilitation sessions using a Numeric-Pain-Rating-Scale (0-10) (NPRS) to evaluate tissue irritability and guide physiotherapy and rehabilitation.
  Use of passive physiotherapy (cold, heat or electric therapies) to treat pain. Active and passive mobilization of the shoulder under the pain threshold, Maitland mobilization, stretch exercises such as: table slides, wall climbers. Use of affected upper limb in pain free Range-of-Motion (ROM) is tolerated and stimulated. Progressively increase time and frequency of Total-End-Range-Time (TERT) positions to increase ROM
  Other Names: Usual care
  Arms: SSNB + IACI
Other: Sham SSNB + IACI — Usual care: All patients complete rehabilitation under supervision of their own physiotherapist. The investigators will provide some guidelines and criteria but is the physiotherapist's choice how to implement these guidelines in clinical practice.
  Patient education on home-exercises Monitoring of peak pain, at rest/night and after rehabilitation sessions using a Numeric-Pain-Rating-Scale (0-10) (NPRS) to evaluate tissue irritability and guide physiotherapy and rehabilitation.
  Use of passive physiotherapy (cold, heat or electric therapies) to treat pain. Active and passive mobilization of the shoulder under the pain threshold, Maitland mobilization, stretch exercises such as: table slides, wall climbers. Use of affected upper limb in pain free Range-of-Motion (ROM) is tolerated and stimulated. Progressively increase time and frequency of Total-End-Range-Time (TERT) positions to increase ROM
  Other Names: Usual care
  Arms: Short-acting SSNB + IACI

SUMMARY:
Frozen shoulder remains a challenging disease to treat as pain and loss of range of motion can persist for many months or even years. This loss of function can have a severe impact on the patient's activities, participation and overall quality of life.

The use of ultrasound-guided (USG) suprascapular nerve blocks (SSNB) and/or intra-articular corticoid injections (IACI) has been supported by many studies. However, double blinded randomized clinical trials using a combination of SSNB and IACI are rare.

The primary objective of this study is to compare the effectiveness of a glenohumeral IACI combined with a SSNB, compared to a glenohumeral IACI combined with a sham SSNB. Outcome measures of interest are shoulder-related disability reported by the patients, shoulder pain and shoulder stiffness. These outcome parameters will be compared between both treatment arms with an intention-to-treat analysis.

As key secondary objectives, the investigators aim to identify which physical examination tests, or combinations of those, are correlated with MRI diagnostic criteria and favor a more positive evolution. Finally, through predictive analysis the investigators will try to establish which patients benefit the most from the combined SSNB + IACI.

DETAILED DESCRIPTION:
Frozen Shoulder (FS) is common disease affecting 2 to 5% of the general population, with a higher prevalence in patients suffering from diabetes and thyroid dysfunction.It remains frustrating for patients and treating health care professionals as severe shoulder pain and loss of function can last for up to two years. 5-7 In the early stage, most patients identify the following symptoms: strong component of night pain, pain with rapid or unguarded movements and aggravated by movement or lying on the affected shoulder.8 Combined with marked pain and limitation in all directions of shoulder range of motion, it is easy to understand that suffering from Frozen Shoulder will have a detrimental effect on quality of life and the ability to perform activities of daily living.

The overall treatment aim for this condition is to "improve pain and function" and treatment goals should be set individually in a shared decision-making process. Patient education on the clinical course and different possible therapeutic interventions, including self-management strategies, should always come first. Clinicians should promote activity modification to utilize pain-free, functional ROM and stretching of the shoulder capsule matching the patient's current level of irritability.

Intra-articular corticosteroid injections (IACI) into the gleno-humeral (GH) joint, combined with shoulder mobility and stretching exercises, have shown to be more effective in providing short-term (4-6weeks) pain relief and improved function compared to exercises alone.

A recent article by Rex et al. places the results of the UK FROST trial in the context of 8 other randomized controlled trials comparing intra-articular corticoid injections (IACI) to manipulation under anesthesia (MUA), arthroscopic capsular release (ACR) and hydrodilatation. These findings did not show clinical superiority of either IACI, MUA nor ACR and evidence for hydrodilatation was inconclusive.

Common sense, in accordance with the National Institute of Health and Care Excellence (NICE) guidelines, recommends that treatments should be offered in a stepped approach from least to most invasive. In their systematic review from 2020, Challoumas et al. show that in the early phase of Frozen Shoulder IA corticosteroid is associated with better short-term outcomes, with possible benefits extending in the mid-terms. These authors recommend to associate IACI to education for home-based exercises and physiotherapy to increase the chances of resolution of symptoms by 6 months.

Unfortunately, not all patients show sufficient improvement in pain and function with IACI and need other therapies. The suprascapular nerve (SSN) provides 60 tot 70% of sensory innervation of the shoulder and suprascapular nerve block (SSNB) has shown in meta-analysis to significantly improve pain and ROM in patients with Frozen Shoulder. This systematic review however has several limitations. Blinding was not always sufficient to rule out a placebo effect, different injections techniques and products (local anesthetics with or without corticosteroids) were used and only data for pain and ROM shoulder could be aggregated as shoulder function was not evaluated in enough trials.

In a rigorous triple blinded RCT, we demonstrated that three successive SSNB with local anesthetics did not improve shoulder pain and function more than three sham injections in patients suffering from subacute Frozen Shoulder. On the other hand, it has been hypothesized that the SSN may be involved in the pathogenesis of Frozen Shoulder and that therefore using optimal approach and drugs (combination of local anesthetics and corticosteroids) in SSNB should be further evaluated in high-quality RCTs.

Evidence suggests that 20mg of triamcinolone or methylprednisolone maybe as effective in frozen shoulder than 40mg but the dosage of 40mg remains most common in clinical and research practice and was chosen to be administered intra-articular in this trial. Trial simulation indicates that the equivalent of 20mg of methylprednisolone is sufficient to increase the mean duration of peripheral nerve blocks and this dosage will be used for SSNB in this study.

In a retrospective review of 102 patients, Jung et al. showed that the combination of an IACI with an SSNB further increased treatment efficacy compared to a single IACI in Frozen Shoulder patients; as pain, ROM and function scored significantly better at different time points (2weeks, 2months and 1 year).

To our knowledge, there has been no previous prospective RCT investigating the added value of an SSNB in combination with an IACI, delivering under ultra-sound guidance the same total amount of corticosteroids in both treatment arms and assuring quadruple blinding (participant, care provider, investigator and outcomes assessor).

The aim of this study is to determine if there is any difference in pain relief and function, as measured by the Shoulder Pain and Disability Index (SPADI), in patients with Frozen Shoulder when given an GH IACI with a SSNB compared to an GH IACI with a sham SSNB. Furthermore, we want to identify which patients will benefit most from GH IACI or the combination of GH IACI and SSNB. The results of this trial will help to guide clinical practice treating patients with FS and improve resource allocation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study must be obtained from the subject prior to initiation of any study-mandated procedure
* Suffering from Frozen Shoulder, defined as: Frozen shoulder is a self-limiting disease characterized by pain and functional restriction in both active and passive shoulder motion lasting more than 1 month, for which radiographic findings of the shoulder joint are unremarkable.
* Dutch or French speaking persons
* Age ≥ 18 years

Exclusion Criteria:

* Subjects with posttraumatic or postsurgical stiff shoulder syndrome
* History of trauma at the onset of symptoms
* Subjects with rheumatologic or neurologic disease involving the shoulder
* Subjects with cervical radiculopathy
* Coagulation disorder
* Hypersensitivity to local anesthetics or MRI contrast agent
* Inability to understand the study procedures
* Psychiatric illness
* Pregnancy
* Subjects who have received prior SSNB in the homolateral shoulder
* Subjects who have received an IACI in the homolateral shoulder in the 3 months before inclusion• Systematic yeast infections
* Hypovolaemia
* Infections at the injection site
* Medical history of malignant hyperthermia, major conduction disorders, acute cardiac decompensation, shock conditions, convulsions

Control subjects for the diagnostic accuracy part of the study protocol

* Inclusion criteria:
* Written informed consent to participate in the study must be obtained from the sub-ject prior to initiation of any study-mandated procedure
* Subjects suffering from shoulder pain that do not fulfill the diagnostic criteria of Frozen Shoulder
* Dutch or French speaking persons
* Age ≥ 18 years
* Contralateral shoulder of Frozen Shoulder subjects
* Exclusion criteria
* Subjects with posttraumatic or postsurgical stiff shoulder syndrome
* History of trauma at the onset of symptoms
* Subjects with rheumatologic or neurologic disease involving the shoulder
* Subjects with cervical radiculopathy
* Coagulation disorder or treatments with anticoagulants
* Hypersensitivity to MRI contrast agent
* Inability to understand the study procedures
* Psychiatric illness
* Pregnancy
* Systematic yeast infections
* Hypovolaemia
* Infections at the injection site
* Medical history of malignant hyperthermia, major conductin disorders, acute cardi-ac decompensation, shock conditions, convulsions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 3 months
  The Shoulder Pain and Disability Index (SPADI) is a self-administered index consisting of 13 items, divided into two subscales: 5 items for pain and 8 items for disability. It can be completed by patients in less than 5 min and has shown good reliability and construct validity in the assessment of shoulder impairments and in particular frozen shoulder. The score for each subscale is obtained by adding up all the individual subscale scores and dividing the result by the maximum subscale score. The normalized score is converted to a scale from 0 to 100, with 100 indicating no problems and 0 indicating serious problems.

SECONDARY OUTCOMES:
Pain - Numeric Pain Rating Scale (NPRS) | 4 weeks - 3 months - 6 months - 12months after the intervention
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). It is the simplest and most commonly used pain rating scale and offers numerous advantages, including ease of administration and scoring, multiple response options, and no reported age-related difficulties in its use.
Shoulder Pain and Disability Index (SPADI) | 4 weeks- 6 months - 12months after the intervention
  The Shoulder Pain and Disability Index (SPADI) is a self-administered index consisting of 13 items, divided into two subscales: 5 items for pain and 8 items for disability. It can be completed by patients in less than 5 min and has shown good reliability and construct validity in the assessment of shoulder impairments and in particular frozen shoulder. The score for each subscale is obtained by adding up all the individual subscale scores and dividing the result by the maximum subscale score. The normalized score is converted to a scale from 0 to 100, with 100 indicating no problems and 0 indicating serious problems.
Constant- Murley score (CMS) | 4weeks - 3 months - 6 months - 12 months after the intervention
  The CMS is a composite scale divided into four sections: pain (15 points), activities of daily living (20 points), ROM (40 points) and strength (25 points) with a total score ranging from 0 (worst possible) to 100 (best possible). Patients were asked to verbally rate each parameter.
Health related quality of life, evaluated with the EuroQol | 4weeks - 3 months - 6 months - 12 months after the intervention
  The EQ-5D 3L is a generic measure of health-related quality of life developed by the EuroQol Group. It is a validated measurement of quality of life widely used in different pathologies. The questionnaire is made up of two parts. The first part is descriptive and uses five different dimensions to score quality of life. These five dimensions are mobility, self-care, activities of the daily life, pain/discomfort and anxiety/depression. There are five different answer possibilities within each dimension, i.e. "no problem", "slight problem", "moderate problem", "severe problem" and "unable to". This renders 3125 different answer possibilities. The second part uses a visual analogue scale (VAS) to score the current health status of the patient, ranging from zero to one hundred. Zero corresponds to death and one hundred corresponds to a (subjective) perfect health status.
PROMIS-29 Upper Extremity v2.0 | 4weeks - 3 months - 6 months - 12 months after the intervention
  The nine-item Patient-Reported Outcomes Measurement Information System (PROMIS)- Upper Extremity short form has been validated against different legacy PROM and general health scores.
  Item-levels are scored numerically for an individual's response to each question.
  PROMIS instruments are always expressed as a score relative to the mean of a group (T-score). The mean score in a population is assigned the value 50. The standard deviation is equal to 10 points. Higher scores (above the mean score) means more of the concept being measured.
Shoulder ROM in abduction, anteflexion, external rotation | 4weeks - 3 months - 6 months - 12 months after the intervention
  Active and passive ROM in anterior elevation, abduction and external rotation are measured using an adapted (large, total length 50cm) goniometer, as described by Riddle et al. and Sabari et al., and values were expressed in degrees °.
Tampa Scale for Kinesiophobia (TSK-11): | 4weeks - 3 months - 6 months - 12 months after the intervention
  A shortened version of the original 17-item TSK, that measures the extent to which a person believes that physical activity or movement may lead to (re)-injury. Patients rate each item on a four-point Likert scale, with scoring alternatives ranging from "strongly disagree" to "strongly agree". Scores range from 11 to 44 with a higher score reflecting greater pain-related fear.
Pain Self-Efficacy Questionnaire (PSEQ) | 4weeks - 3months - 6 months - 12 months after the intervention
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item scale which assesses a person's confidence in the ability to perform a task or activity, despite the pain. Each item is scored on a seven-point Likert scale (from "not at all confident" to "completely confident"). The total score ranges from 0 to 60 with a higher score representing greater pain self-efficacy beliefs.
Global Rating of Change Score (GRoC) | 4weeks - 3months - 6 months - 12 months after the intervention
  The Global Rating of Change Score (GRoC) is a frequently used outcome measure that is used independently to measure improvements in a patient's condition or as an anchor for other outcomes measures. On 11-point Likert scale participants rate the clinical course of their condition since the start of the treatment: from -5 "a great deal worse" to +5 "a great deal better" with 0 being "no change".
Work Ability Index (WAI) | 4weeks - 3months - 6 months - 12 months after the intervention
  The Work Ability Index (WAI) measures the work ability considering physical and mental parts of work as well as different diseases and their impact on work ability. It's a 10 items questionnaire concerning current work ability compared with the lifetime best, work ability in relation to the job demands, number of current diseases diagnosed by a physician, estimated work impairment due to diseases, sick leave, self-prognosis of work ability and mental resources.
  A given answer to a question earns points. The sum of all these points results in the WAI score, which ranges from 7 to 49 points. The score indicates the extent to which the individual's capabilities and the job requirements are consistent with each other, a higher score indicating a better match between capabilities and job requirements.
Work Status | 4weeks - 3months - 6 months - 12 months after the intervention
  Work status: Health economic assessment: As the investigators expect subgroups of Frozen Shoulder to be unable to work, subjects will be questioned if they are incapacitated to work due to Frozen Shoulder during baseline assessments. Once the symptoms and function improve, the investigators expect patients to be able to return to work.
Health care service use | 4weeks - 3months - 6 months - 12 months after the intervention
  Patients will keep a diary to log usage of pain medication and physiotherapy visits
Adverse effects | 4weeks - 3months - 6 months - 12 months after the intervention
  At every patient study contact, the occurrence or not of adverse affects will be recorded.
Rescue therapy | 3months - 6months - 12months after the intervention
  As this is a pragmatic trial, patients will be offered rescue therapy, consisting of an USG SSNB + IACI in their affected shoulder, every 3 months after inclusion, with a maximum of 3 interventions in 12 months

OTHER OUTCOMES:
Superiority analysis of shoulder-related disability, pain and shoulder stiffness at 6 months after start of enrolment. | 6 months after start of enrolment
  An intermediary statistical analysis will be performed at 6 months after start of enrolment. In case all 3 outcomes (disability, pain, shoulder stiffness) show non-superiority at 6m, the study will not be extended to the 12-month time point.
Exploratory prediction analysis: part 1 | 18 months after inclusion
  Through regression analysis the investigators want to find out which factors predict I) SPADI score at 3 -6- 12 months follow-up, II) pain NPR level at 3-6-12 months, III) shoulder ROM (°) at 3-6-12 months and IV) return to work and WAI score at 3-6-12 months.
  The initial set of predictor variables, baseline values, that will be considered is :
  1. SPADI score
  2. Presence of joint capsule enhancement on MRI: (yes/no)
  3. Shoulder ROM (°)
  4. Age (years)
  5. Gender (male/female)
  5. Duration of symptoms to intervention (weeks) 6. Presence of diabetes (yes/no)
Exploratory prediction analysis: part 2 | 18 months after inclusion
  Through regression analysis the investigators want to identify which physical examination tests, or which combinations of tests are correlated with MRI diagnostic criteria and a more positive evolution of SPADI score - NPR pain score - shoulder ROM (°)- Return to Work (RTW)/WAI score:
  The initial set of predictor variables, baseline values, that will be considered is :
  1. SPADI score
  2. Presence of joint capsule enhancement on MRI: (yes/no)
  3. Shoulder ROM (°)
  4. Age (years)
  5. Gender (male/female)
  5. Duration of symptoms to intervention (weeks) 6. Presence of diabetes (yes/no)
Exploratory prediction analysis: part 3 | 18 months after inclusion
  Through regression analysis the investigators want to identify patients that benefit the most from the combined SSNB + IACI
  The initial set of predictor variables, baseline values, that will be considered is :
  1. SPADI score
  2. Presence of joint capsule enhancement on MRI: (yes/no)
  3. Shoulder ROM (°)
  4. Age (years)
  5. Gender (male/female)
  5. Duration of symptoms to intervention (weeks) 6. Presence of diabetes (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schiltz, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Data will be published in peer review journal on completion of the study.

REFERENCES:
- [Background] Schiltz M, Goudman L, Moens M, Nijs J, Hatem SM. The diagnostic value of physical examination tests in adhesive capsulitis: a systematic review. Eur J Phys Rehabil Med. 2023 Dec;59(6):724-730. doi: 10.23736/S1973-9087.23.07940-6. Epub 2023 Sep 22. PMID 37737049
- [Background] Jump CM, Waghmare A, Mati W, Malik RA, Charalambous CP. The Impact of Suprascapular Nerve Interventions in Patients with Frozen Shoulder: A Systematic Review and Meta-Analysis. JBJS Rev. 2021 Dec 22;9(12). doi: 10.2106/JBJS.RVW.21.00042. PMID 34936584
- [Background] Kelley MJ, Shaffer MA, Kuhn JE, Michener LA, Seitz AL, Uhl TL, Godges JJ, McClure PW. Shoulder pain and mobility deficits: adhesive capsulitis. J Orthop Sports Phys Ther. 2013 May;43(5):A1-31. doi: 10.2519/jospt.2013.0302. Epub 2013 Apr 30. No abstract available. PMID 23636125
- [Background] Millar NL, Meakins A, Struyf F, Willmore E, Campbell AL, Kirwan PD, Akbar M, Moore L, Ronquillo JC, Murrell GAC, Rodeo SA. Frozen shoulder. Nat Rev Dis Primers. 2022 Sep 8;8(1):59. doi: 10.1038/s41572-022-00386-2. PMID 36075904
- [Derived] Schiltz M, Croes J, van Brabander L, Roggeman S, Goudman L, Moens M, Nijs J, Pouliart N, Forthomme B, Hatem SM. The FROSTBLOCK trial: Protocol for a randomized controlled trial of intra-articular corticosteroid injection with or without suprascapular nerve block in frozen shoulder. Trials. 2025 Sep 29;26(1):383. doi: 10.1186/s13063-025-09123-y. PMID 41023761